CLINICAL TRIAL: NCT02439996
Title: Different Doses of IVIG for Kawasaki Disease: a Multicentre, Prospective, Randomised Trial
Brief Title: Different Doses of IVIG for Kawasaki Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Children's Medical Center (Other); Shanghai Children's Hospital (Other)
Responsible Party: Principal Investigator, Guoying huang, Professor,President, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KD(2015-2016)
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Kawasaki Disease
Keywords: Kawasaki disease IVIG
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Immunoglobulins, Intravenous; acetylsalicylic acid lysinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IVIG(1g/kg,once) (Experimental): The KD children will be randomly assigned to three groups. The patients in group C will receive IVIG 1g/kg once.
  Interventions: Drug: IVIG (1g/kg,once)
- IVIG(1g/kg,twice) (Experimental): The KD children will be randomly assigned to three groups. The patients in group B will receive IVIG 1g/kg for 2 days continuousl.
  Interventions: Drug: IVIG (1g/kg,twice)
- IVIG(2g/kg.once) (Active Comparator): The KD children will be randomly assigned to three groups. The patients in group A will receive IVIG 2g/kg once.
  Interventions: Drug: IVIG (2g/kg.once)

INTERVENTIONS:
Drug: IVIG (1g/kg,once) — Group C patients received IVIG 1g/kg per day once. The IVIG was started on the fifth to tenth day of illness. In combination with IVIG, the patients were administered aspirin at a dose of 30 mg/kg per day; this dose was reduced to 3-5 mg/kg per day after the fever disappeared for 3 days and the CRP value was ≤8mg/L. Patients who were admitted before the fourth day of illness were treated only with aspirin. Each immunoglobulin was administered at a dose of 1 g/kg for 10h.
  Patients who did not respond to initial IVIG therapy were given a second dose of IVIG 24-36 hours after the initial dose at 2g/kg. Patients who did not respond to second dose IVIG were given methylprednisolone 10mg/kg for 3 days or infliximab 5mg/kg once.
  Other Names: Asprin
  Arms: IVIG(1g/kg,once)
Drug: IVIG (1g/kg,twice) — Group B patients received IVIG 1g/kg for 2 days continuously. The IVIG was started on the fifth to tenth day of illness. In combination with IVIG, the patients were administered aspirin at a dose of 30 mg/kg per day; this dose was reduced to 3-5 mg/kg per day after the fever disappeared for 3 days and the CRP value was ≤8mg/L. Patients who were admitted before the fourth day of illness were treated only with aspirin. Each immunoglobulin was administered at a dose of 1 g/kg for 10h.
  Patients who did not respond to initial IVIG therapy were given a second dose of IVIG 24-36 hours after the initial dose at 2g/kg. Patients who did not respond to second dose IVIG were given methylprednisolone 10mg/kg for 3 days or infliximab 5mg/kg once.
  Other Names: Asprin
  Arms: IVIG(1g/kg,twice)
Drug: IVIG (2g/kg.once) — Group A patients received IVIG 2g/kg per day once. The IVIG was started on the fifth to tenth day of illness. In combination with IVIG, the patients were administered aspirin at a dose of 30 mg/kg per day; this dose was reduced to 3-5 mg/kg per day after the fever disappeared for 3 days and the CRP value was ≤8mg/L. Patients who were admitted before the fourth day of illness were treated only with aspirin. Each immunoglobulin was administered at a dose of 1 g/kg for 10h.
  Patients who did not respond to initial IVIG therapy were given a second dose of IVIG 24-36 hours after the initial dose at 2g/kg. Patients who did not respond to second dose IVIG were given methylprednisolone 10mg/kg for 3 days or infliximab 5mg/kg once.
  Other Names: Asprin
  Arms: IVIG(2g/kg.once)

SUMMARY:
The objective of this study is to investigate the effect of different doses of intravenous immunoglobulin (IVIG) (1g/kg once, 1g/kg twice, 2g/kg once) for Kawasaki disease (KD) in a multicentre, prospective,randomised trial.

DETAILED DESCRIPTION:
Kawasaki disease is an acute febrile illness recognized most often in young children. Coronary abnormality is the most serious complication preventable with intravenous immunoglobulin (IVIG) administration. Various treatment regimens of IVIG have been reported.The optimal administrative doses of IVIG deserves more observations.We will conduct a multicenter, randomized, prospective trial to determine the effect of different doses of IVIG (1g/kg once, 1g/kg twice, 2g/kg once) for Kawasaki disease. The KD children will be randomly assigned to three groups and were given different IVIG regimen (1g/kg once, 1g/kg twice, 2g/kg once)as initial treatment. Patient age, gender, white blood cell count, hemoglobin, erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), red blood cell specific volume (HCT) , serum albumin, the fever days,and the cost of hospital stay will be analyzed among the three groups. The primary outcome is the duration of fever subsided and the incidence of coronary artery lesions .

ELIGIBILITY:
Inclusion Criteria:

* Individual patient's medical file data confirmed the diagnosis of KD using the 5th revised edition of diagnostic criteria for KD, issued by the Japan Kawasaki Disease Research Committee at the 7th International Kawasaki Disease Symposium in 2002.
* the patients aged from 1 months to 12 years old.
* All included patients required to sign an informed consent form.
* the patients didn't receive treatment before.

Exclusion Criteria:

* The patients with the application of hormone or other immunosuppressive agents;
* The patients didn't want to signed informed consent.

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 404 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Duration of fever subsided to normal after initial IVIG finished | 36 hours after IVIG finished
  Hours of fever subsided to normal after initial IVIG finished
incidence of coronary artery lesions(CAL) after IVIG finished | start from IVIG finished, ended by the end of 2 weeks
  incidence of coronary artery lesions(CAL) after IVIG finished diagnosed by echocardiography

SECONDARY OUTCOMES:
incidence of coronary artery lesions(CAL) after IVIG finished | start from IVIG finished, ended by the end of 1 month
  incidence of coronary artery lesions(CAL) after IVIG finished diagnosed by echocardiography
incidence of coronary artery lesions(CAL) after IVIG finished | start from IVIG finished, ended by the end of 3 month
  incidence of coronary artery lesions(CAL) after IVIG finished diagnosed by echocardiography
incidence of coronary artery lesions(CAL) after IVIG finished | start from IVIG finished, ended by the end of 6 month
  incidence of coronary artery lesions(CAL) after IVIG finished diagnosed by echocardiography and coronary atery angiogram
Total dose of immunoglobin used for every patient | estimated about up to 10 days, start from admission,ended by discharge
  Total dose of immunoglobin used for every patient
total medical cost for KD treatment during hospital stay | estimated about up to 10 days, start from admission,ended by discharge
  record the hospital duration of every patient and the medical expenses for KD
total frequency (%) of severe adverse events | estimated about up to 10 days, start from admission,ended by discharge
  Severe adverse events included death, infection or exacerbation, heart failure, allergic reaction, etc

CONTACTS AND LOCATIONS:
Overall Officials: Guoying Huang, PHD, Study Chair — Children Hospital of Fudan University
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] He L, Liu F, Yan W, Huang M, Huang M, Xie L, Guo Y, Xu X, Chu C, Wu L, Liang X, Sun S, Wang F, Zhao L, Zhao Q, Ma X, Xie L, Huang G. Randomized trial of different initial intravenous immunoglobulin regimens in Kawasaki disease. Pediatr Int. 2021 Jul;63(7):757-763. doi: 10.1111/ped.14656. Epub 2021 Jun 16. PMID 33600060